CLINICAL TRIAL: NCT02307370
Title: Atherectomy By Laser Ablation With Turbo-Elite
Acronym: ABLATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D024204
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Turbo-Elite Atherectomy (Experimental)
  Interventions: Device: Turbo-Elite Laser Catheter

INTERVENTIONS:
Device: Turbo-Elite Laser Catheter — Application of laser energy to remove blockage

SUMMARY:
The primary objective for this study is to prove the safety and effectiveness of the Spectranetics Turbo-Elite catheter in atherectomy treatment for infrainguinal arteries with catheter to vessel sizing of at least 50%.

ELIGIBILITY:
Inclusion Criteria:

* PAD with Rutherford Class 1-4
* Patient is able to walk unassisted or with non-motorized assistive devices.
* Documented PAD by ABI <0.9 or previous intervention with reoccurrence of symptoms
* Documented stenosis by duplex ≥50%

Exclusion Criteria:

* Patient is pregnant or breast feeding.
* Evidence of Acute Limb Ischemia within 7 days prior to procedure.
* CVA < 60 days prior to procedure.
* MI < 60 days prior to procedure.
* Known contraindication to aspirin, antiplatelet/anti-coagulant therapies required for procedure/follow up.
* Known allergy to contrast media that cannot adequately be pre-medicated prior to study procedure.
* Uncontrolled hypercoagulability or history of HIT or HITTS syndrome.
* Serum creatinine ≥ 2.5 mg/dL (unless dialysis-dependent) within one day prior to procedure.
* Patient is simultaneously participating in another investigational drug or device study that will interfere with the 30 day Safety Endpoint.
* Previously identified severe calcium in the vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Turbo-Elite Atherectomy
Started | 44
30 Day Follow-up | 40
180 Day Patient Telephone Contact | 25
Completed | 25
Not Completed | 19
Not completed — Death | 5
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Declined Addendum ICF | 6
Not completed — No response during telephone contact | 5
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: One study center enrolled only one study participant, but due to site compliance, data was never collected for the study. This study center was closed due to the non-compliance issue. As a result, 44 participants were enrolled but data is available only for 43 participants.
Arm/Group | Turbo-Elite Atherectomy
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Weight (kg) [Mean (Standard Deviation); unit: kg] | 82.8 (20.6)
Height (cm) [Mean (Standard Deviation); unit: cm] | 168.0 (9.1)
Medical History [Count of Participants; unit: Participants]
  History of Hypertension | 39
  History of Hyperlipidemia | 40
  History of Diabetes Mellitus | 21
  History of Coronary Artery Disease | 26
  History of Cebrovascular Accident | 2
Smoking Status [Count of Participants; unit: Participants]
  Never | 8
  Current | 9
  Stopped | 26

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint - Mean Reduction in Percent Stenosis
Description: The primary efficacy endpoint target was a mean reduction in percent stenosis of greater than 20% in each study participating at the time of the procedure by Angiographic Core Lab assessment after Turbo-Elite use. A participant showing a mean reduction of 20% was considered a success for the primary efficacy endpoint.
Time Frame: Day 1
Population: The analysis set is composed of 43 patients, data for primary efficacy analysis was available only for 42 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Turbo-Elite Atherectomy
Number analyzed (Participants) | 42
Participants | 39

2. Primary Outcome: Primary Safety Endpoint is Freedom From Major Adverse Event (MAE)
Description: The primary safety endpoint target was 80% of study participant with freedom from a Major Adverse Event (MAE) through 30 day follow-up. A MAE was defined as: all cause death, major amputation in the target limb, or target lesion revascularization.
Time Frame: 30 day follow-up
Population: Although 40 participants completed 30 day follow-up, data was only available for 39 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Turbo-Elite Atherectomy
Number analyzed (Participants) | 39
Participants | 38

3. Secondary Outcome: Final Procedure Residual Stenosis After All Therapy
Description: A Final Procedure Residual Stenosis by visual assessment after all therapy will be accessed acutely during the procedure.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Final Residual Stenosis % Per Site
Arm/Group | Turbo-Elite Atherectomy
Number analyzed (Participants) | 43
Final Residual Stenosis % Per Site | 12.7 (13.1)

4. Secondary Outcome: Characterization of Adjunctive Therapy Use
Description: Adjunctive therapy use will be characterized by frequencies.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Turbo-Elite Atherectomy
Number analyzed (Participants) | 43
Participants
  Turbo-Tandem (atherectomy laser) | 0
  Standard Balloon Angioplasty | 23
  Drug Coated Balloon Angioplasty | 20
  Stenting | 14

5. Secondary Outcome: Ankle-Brachial Index (ABI) Change From Baseline to 30 Days.
Description: ABI will be assessed at baseline and within 30 days of the procedure. The ABI is calculated ratio of the highest ankle blood pressure to the highest arm blood pressure. The ABI is a non-invasive tool for screening for Peripheral Artery Disease.
Time Frame: Baseline and 30 Days post-procedure
Population: Although 43 patients were part of the analysis set, ABI is one of the most often missed assessments during baseline and the follow-up period. Only 40 participants had available ABI data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Turbo-Elite Atherectomy
Number analyzed (Participants) | 40
ratio
  Screening | 0.7 (0.2)
  30-day | 0.9 (0.3)
  Change from Screening to 30 days | 0.3 (0.3)

6. Secondary Outcome: Rutherford Class (RCC) Change
Description: Rutherford Class (RCC) will be assessed at baseline and within 30 days of the procedure. The Rutherford-Becker Clinical Categories (RCC) are a classification system of chronic limb ischemia ranging from 0 (asymptomatic; no hemodynamically significant occlusive disease) to 6 (major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable). Lower categories represent better clinical status.
Time Frame: Baseline and 30 days of procedure
Population: Refer to participant flow.
Measure: Count of Participants; unit: Participants
Groups:
- Turbo-Elite Atherectomy (Screening); Turbo-Elite Atherectomy (30-day Follow-up): Turbo-Elite Laser Catheter: Application of laser energy to remove blockage
Arm/Group | Turbo-Elite Atherectomy (Screening) | Turbo-Elite Atherectomy (30-day Follow-up)
Number analyzed (Participants) | 43 | 40
Participants
  Rutherford Class 0 | 0 | 17
  Rutherford Class 1 | 0 | 11
  Rutherford Class 2 | 2 | 5
  Rutherford Class 3 | 33 | 7
  Rutherford Class 4 | 8 | 0
  Rutherford Class 5 | 0 | 0
  Rutherford Class 6 | 0 | 0

7. Secondary Outcome: Freedom From Target Lesion Revascularization (TLR) Through 180 Days.
Description: Freedom from target lesion revascularization (TLR) through 180 days post procedure
Time Frame: Day 180 (6 Months)
Measure: Count of Participants; unit: Participants
Arm/Group | Turbo-Elite Atherectomy
Number analyzed (Participants) | 43
Participants | 40

ADVERSE EVENTS:
Arm/Group | Turbo-Elite Atherectomy
All-Cause Mortality (participants affected / at risk) | 5/43
Serious Adverse Events (participants affected / at risk) | 14/43
Other Adverse Events (participants affected / at risk) | 2/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turbo-Elite Atherectomy (N=43)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Arterial Dissection (Vascular disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Restenosis - Target Lesion (Vascular disorders) | 3 (3)
Restenosis - Target Vessel (Vascular disorders) | 1 (1)
Restenosis - Non-Target Limb (Vascular disorders) | 5 (5)
Restenosis - Non-Target Vessel (Vascular disorders) | 1 (1)
Stroke (Cardiac disorders) | 1 (1)
Other - Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Other - Cardiac (Cardiac disorders) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turbo-Elite Atherectomy (N=43)
Arterial Perforation (Vascular disorders) | 1 (1)
Embolism (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No